CLINICAL TRIAL: NCT00050349
Title: EPO906 Therapy in Patients With Metastatic Carcinoid Tumors and Other Neuroendocrine Tumors
Brief Title: EPO906 in Carcinoid and Other Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2212
Record Dates: First submitted 2002-12-04; First posted 2002-12-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2013-03

CONDITIONS: Carcinoid; Neuroendocrine Tumors
Keywords: cancer; tumor; tumour; neoplasm; carcinoma; carcinoid; neuroendocrine; Islet cell; Gastrinoma; VIPoma; metastatic; intravenous; epothilone
MeSH Terms: conditions — Carcinoid Tumor; Neuroendocrine Tumors; Neoplasms; Carcinoma; Gastrinoma; Vipoma; Neoplasm Metastasis | interventions — epothilone B

ARMS (1):
- EPO906 (Experimental)
  Interventions: Drug: EPO906 epothilone B

INTERVENTIONS:
Drug: EPO906 epothilone B
  Other Names: patupilone

SUMMARY:
This study will examine whether the new investigational drug EPO906, given by intravenous infusion (IV directly into the vein), is effective in shrinking tumors and preventing the growth of cells that cause metastatic carcinoid and other neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven metastatic carcinoid tumors or other neuroendocrine tumors (Islet cell, Gastrinomas and VIPomas) with at least one measurable lesion (other than bone) that has either not been previously irradiated or if previously irradiated has demonstrated progression since the radiation therapy
* The patient has no major impairment of renal or hepatic function, as defined by the following laboratory parameters: total bilirubin <1.5 X ULN; AST, ALT<2.5X ULN (<5 X ULN if liver metastases are present)
* Patients on Sandostatin Lar (long acting somatostatin analogue) must be on a stable dose for 30 days prior to study entry and short acting somatostatin analogues must be judged to be on a clinically stable dose by the investigator prior to study entry
* Must have a life expectancy of greater than three (3) months
* Karnofsky Performance Status > 60
* Female patients must have a negative serum pregnancy test at screening. (Not applicable to patients with bilateral oophorectomy and/or hysterectomy or to those patients who are postmenopausal.)

Exclusion Criteria:

* Patients with symptomatic CNS metastases or leptomeningeal involvement
* Patients with known brain metastases, unless these metastases have been treated and/or have been stable for at least six months prior to study start. Subjects with a history of brain metastases must have a head CT with contrast to document either response or progression.
* Patients with bone metastases as the only site(s) of measurable disease
* Patients with hepatic artery chemoembolization within the last 6 months (one month if there are other sites of measurable disease)
* Patients who have been previously treated with radioactive directed therapies
* Patients who have been previously treated with epothilone
* Patients with any peripheral neuropathy or unresolved diarrhea greater than Grade 1
* Patients with severe cardiac insufficiency patients taking Coumadin or other warfarin-containing agents with the exception of low dose warfarin (1 mg or less) for the maintenance of in-dwelling lines or ports
* Patients taking any experimental therapies history of another malignancy within 5 years prior to study entry except curatively treated non-melanoma skin cancer, prostate cancer, or cervical cancer in situ
* Patients with active or suspected acute or chronic uncontrolled infection including abcesses or fistulae
* Patients with a medical or psychiatric illness that would preclude study or informed consent and/or history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits
* HIV+ patients
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Tumor response as assessed by radiologic techniques and/or physical examination based on Response Evaluation Criteria in Solid Tumors (RECIST) | every 12 weeks

SECONDARY OUTCOMES:
Time to progression | until documented disease progression, death or date of follow up
Overall survival | after treatment, every 3 months (maximum of 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - LSU HEALTH SCIENCES CENTER/ LSU SCHOOL OF MEDICINE Deptof LSU Health Sciences (2), New Orleans, Louisiana
  - Weill Medical College of Cornell Univ., New York, New York
  - Oregon Health Sciences University, Portland, Oregon